CLINICAL TRIAL: NCT07263113
Title: Evaluation of the Association Between the Effects of Generalized Stage 3 and 4 Periodontitis on Arterial Stiffness and Cardiovascular Risk: the PAROCAR Study
Acronym: PAROCAR
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Nantes University Hospital (Other)
Collaborators: French Interregional Group of Clinical Research and Innovation (Other); Université de Nantes (Other); Axelife company (Unknown)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: RC25_0304; 2025-A01525-44 (Other: ANSM)
Record Dates: First submitted 2025-11-21; First posted 2025-12-04 (Actual); Last update posted 2025-12-04 (Actual); Status verified 2025-12

CONDITIONS: Periodontis; Atherosclerosis Cardiovascular Disease
Keywords: periodontis; Atherosclerosis; Cardiovascular Risk; Arterial Stiffness
MeSH Terms: conditions — Atherosclerosis

STUDY DESIGN:
Intervention Model Description: Parallel observational groups
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Exposed group (periodontitis) (Other): Patients diagnosed with generalized stage 3 or 4 periodontitis (Chicago 2017 Classification).
  Interventions: Other: Periodontal examination and pulse wave velocity
- Non-exposed group (healthy control) (Other): Patients with a healthy periodontium and no history of periodontal disease.
  Interventions: Other: Periodontal examination and pulse wave velocity

INTERVENTIONS:
Other: Periodontal examination and pulse wave velocity — Clinical oral examination (plaque index, bleeding on probing, probing depth, clinical attachment loss), lipid profile measurement, anthropometric and hemodynamic assessments (BMI, blood pressure, pulse wave velocity).

SUMMARY:
Periodontal diseases are chronic inflammatory conditions affecting nearly half of the adult population and are associated with systemic inflammatory responses. Recent evidence suggests a possible link between severe periodontitis and cardiovascular diseases through shared inflammatory pathways.

The PAROCAR study aims to evaluate the association between generalized periodontitis (stages 3 and 4, 2017 Chicago Classification) and arterial stiffness measured by pulse wave velocity (PWV), compared to matched controls without periodontitis, adjusted for conventional cardiovascular risk factors.

DETAILED DESCRIPTION:
Periodontal disease is the sixth most prevalent human disease, affecting 45-50% of the adult population, with 11.2% exhibiting severe forms (stages 3 and 4). This chronic inflammation of the gingiva, caused by dysbiosis of the subgingival microbiota, leads to progressive destruction of the supporting tissues of the teeth (alveolar bone and periodontal ligament) and induces local and systemic inflammatory responses.

The translocation of periodontal bacteria and their metabolites into the bloodstream, as well as the systemic release of inflammatory mediators such as C-reactive protein (CRP), interleukins (IL-1β, IL-6), and tumor necrosis factor-alpha (TNF-α), contributes to endothelial dysfunction and oxidative stress. These mechanisms are thought to play a role in the initiation and progression of atherosclerotic lesions, thus linking periodontitis to cardiovascular disease development.

The PAROCAR study aims to provide a proof of concept of the contributory role of severe periodontitis in cardiovascular risk by comparing arterial stiffness between subjects with generalized periodontitis (stage 3-4) and healthy controls.

This is a monocentric, prospective, cross-sectional, observational, exposed/non-exposed study conducted at the Dental Care Center of Nantes University Hospital.

A total of 206 participants will be included:

* 103 exposed subjects with generalized stage 3-4 periodontitis, diagnosed according to the 2017 Chicago Classification
* 103 non-exposed healthy controls, with no clinical or radiographic signs of periodontal disease.

Participants will be strictly matched according to their cardiovascular risk profile, using the SCORE2 algorithm recommended by the European Society of Cardiology (ESC, 2021). SCORE2 estimates the 10-year risk of a first fatal or non-fatal atherosclerotic cardiovascular event based on age, sex, systolic blood pressure, total cholesterol, HDL cholesterol, and smoking status.

Matching by SCORE2 ensures that both groups (periodontitis and control) have equivalent baseline cardiovascular risk levels, thereby minimizing the influence of classical confounders such as age, sex, lipid levels, or hypertension. This approach isolates the potential intrinsic contribution of periodontal inflammation to increased arterial stiffness.

The primary endpoint is the comparison of the mean pulse wave velocity (PWV) between exposed and non-exposed groups.

The secondary endpoints are the correlations between PWV and periodontal severity indices (plaque index, bleeding on probing, probing depth, clinical attachment loss, and staging/grading).

Anthropometric and hemodynamic parameters (BMI, blood pressure, lipid profile) will also be collected to control for potential confounding factors.

By clarifying whether severe periodontitis independently affects arterial stiffness, the PAROCAR study may help refine cardiovascular risk stratification tools and open new perspectives for preventive strategies integrating oral health into global cardiovascular prevention policies

ELIGIBILITY:
Inclusion Criteria:

* Age 40-69 years
* Minimum of 12 teeth (3 per quadrant)
* Written informed consent Exposed group: generalized periodontitis stage 3 or 4 (Chicago 2017 Classification) Non-exposed group: healthy periodontium

Exclusion Criteria:

* Patients diagnosed with diabetes,
* Patients diagnosed with hypertension or with a history of severe cardiovascular disease,
* Patients diagnosed with familial hypercholesterolaemia,
* Patients with a medical history or current condition that, in the investigator's opinion, is likely to interfere with the study results,
* Patients with a BMI ≥ 30 kg/m²,
* Patients who have previously undergone periodontal treatment,
* Patients who consume more than 2 units of alcohol per day,
* Patients who refuse to participate in the study,
* Minors and patients under the age of 40,
* Adult patients under legal protection (guardianship, curatorship),
* Patients deprived of their liberty,
* Pregnant or breastfeeding women,
* Patients not affiliated with a health insurance scheme (AME)
* Patients already included in another interventional study

Ages: 40 Years to 69 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 206 (Estimated)
Dates: Start 2025-12-01 (Estimated); Primary Completion 2027-12-01 (Estimated); Study Completion 2027-12-01 (Estimated)

PRIMARY OUTCOMES:
Difference in mean pulse wave velocity between exposed and non-exposed groups. | Day 1 At the single study visit
  Comparison of the mean pulse wave velocity (PWV) values between patients with generalized periodontitis and healthy controls, using a Class IIa medical device (pOpmètre®) based on photoplethysmography technology.

SECONDARY OUTCOMES:
Correlation between periodontitis severity (stage 3 or stage 4) and pulse wave velocity. | Day 1 At the single study visit
  Assessment of the correlation between arterial stiffness, measured by pulse wave velocity (PWV), and the severity of periodontitis evaluated through periodontal health indicators, including dental plaque accumulation (O'Leary index), bleeding on probing, pocket depth, gingival recession, and clinical attachment loss, as defined by the 2017 Chicago Classification.